CLINICAL TRIAL: NCT02377778
Title: Comparative Effect of Theipoental and Propofol in IVF Outcome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHR-8
Record Dates: First submitted 2015-02-25; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — Propofol; Thiopental

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Experimental): In this arm patients will be receiving propofol for anaesthesia at doses 3-5mg depending on the time needed to complete oocyte retrieval
  Interventions: Drug: Propofol
- Thiopental (Active Comparator): In this arm patients will receive thiopental for anaesthesia at doses 7mg and a repeat dose of 2-3mg depending on the time needed to completed oocyte retrieval
  Interventions: Drug: Thiopental

INTERVENTIONS:
Drug: Propofol — Propofol intravenous infusion for introduction and maintance of anaesthesia at doses 3-5mg depending on the total time needed for completion of oocyte retrieval
  Arms: Propofol
Drug: Thiopental — Patients will receive thiopental in addition to fentanyl for introduction and maintanance of anaesthesia at doses 7mg. IF required patients will receive a repeat dose of 1-3mg of thiopental depending on the totla time needed to complete oocyte retrieval
  Arms: Thiopental

SUMMARY:
In this study the aim is to compare the effect of the type of anaesthetic drug used during oocyte retrieval on fertilization rates of oocytes retrieved after ovarian stimulation for in-vitro fertilization.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing oocyte retrieval for IVF under general anesthesia
* age ≤45 years

Exclusion Criteria:

* women with a known hypersensitivity to the active substance of the investigating drugs or any of their excipients

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | First 24h after oocyte retrieval
  The number of oocytes fertilized divided by the number of oocytes in which fertilization was attempted per randomized patient

SECONDARY OUTCOMES:
Number of MII oocytes | 12h after oocyte rertieval
Pregnancy rate | 14 days after embryo transfer
  Patients with positive (>20 IU/L) b-hCG test at 14 days after embryo transfer
Implantation rate | 40 days after embryo traansfer
  Number of gestational sacs per embryos transferred per patient
The concentration of propofol or thiopental in the follicular fluid of the dominant (larger) follicle aspirated at oocyte retrieval | 12 hours after oocyte retrieval

CONTACTS AND LOCATIONS:
Locations (1):
- Unit for Human Reproduction, 1st Dept of OB/Gyn, Medical School, Aristotle UNiversity of Thessaloniki, Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Goutziomitrou E, Venetis CA, Kolibianakis EM, Bosdou JK, Parlapani A, Grimbizis G, Tarlatzis BC. Propofol versus thiopental sodium as anaesthetic agents for oocyte retrieval: a randomized controlled trial. Reprod Biomed Online. 2015 Dec;31(6):752-9. doi: 10.1016/j.rbmo.2015.08.013. Epub 2015 Sep 4. PMID 26515147